CLINICAL TRIAL: NCT02518360
Title: Effect of Osteopathic Treatment in Patients With Nonspecific Low Back Pain: Stabilometry
Brief Title: Osteopathic Treatment in Patients With Low Back Pain: Stabilometry
Acronym: Osteop-COP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Emilio-José Poveda-Pagán, PT - PhD, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversidadMHE
Record Dates: First submitted 2015-08-02; First posted 2015-08-07 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Lower Back Pain
Keywords: NON SPECIFIC LOW BACK PAIN; OSTEOPATHY; FOOT PRESSURE PLATFORM; POSTURAL BALANCE
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSTEOPATHIC PROTOCOL (Experimental): Physiotherapist applies an osteopathic treatment in non-specific low back pain patients.
  The experimental group is treated with osteopathy, three sessions (20 minutes/session) and a frequency one session/week. Osteopathic treatment osteopathic is a body adjustment protocol. This protocol adjusts the musculoskeletal disorders since neck to lower limbs in the experimental group. Before treatment, immediately after the last session and a month later, are measured stabilometric parameters, height and Oswestry.
  Interventions: Other: Osteopathic
- Auto Stretching (Active Comparator): The patients realizes stretching protocol: two stretching global postures once a week (10 minutes for each posture) for three weeks: the first is for the anterior muscular chain and the second posture to stretch the posterior muscle chain. Before three stretching, immediately after the last session and a month later, are measured stabilometric parameters, height and Oswestry.
  Interventions: Other: Auto Stretching

INTERVENTIONS:
Other: Osteopathic — Body adjustment in three sessions (20 minutes/session).
  Other Names: Manual Therapy; Muscle chains
  Arms: OSTEOPATHIC PROTOCOL
Other: Auto Stretching — The patients realize auto stretching in three sessions (20 minutes/session).
  Other Names: Muscle chains
  Arms: Auto Stretching

SUMMARY:
Determine the improvement in nonspecific low back pain patients with osteopathic techniques (Body Adjustment Protocol) and know changes in stabilometric measures analyzed with a stabilometric platform (Footscan®).

DETAILED DESCRIPTION:
Fifty patients participate in this study (25 experimental group with body adjustment protocol of osteopathy and 25 control group). For a first objective of this study, all the patients determine if the osteopathic approach to the body adjustment approach will improve low back pain (Oswestry Questionnaire). For the second aim, the investigators want to know if there are changes in the distribution of body weight in lower limbs in group experimental and control group, analyzed with a stabilometric platform (Footscan®).

The experimental group is treated with osteopathy, three sessions (20 minutes/session) and a frequency one session/week. The treatment osteopathic is the body adjustment protocol. In the other hand, the control group made 2 stretching global postures once a week (10 minutes for each posture) for three weeks: the first was for the anterior muscular chain and the second posture to stretch the posterior muscle chain. Before treatment, immediately after the last session and a month later, are measured stabilometric parameters, height and Oswestry.

The analysis will be made with Statistical Package for the Social Sciences (SPSS Statistics) 22.0

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Patients with non-specific low back pain.
* Patients with alteration in the distribution of loads in a podiatric platform.

Exclusion Criteria:

* Specific low back pain diagnosed.
* Pregnancy.
* Recent surgery in the last year.
* Acute musculoskeletal disorders out of the lumbar region.
* Patients with vestibular and instability problems.
* Meniere syndrome.
* Oncologic patients.
* Patients with manual therapy treatment during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Oswestry Questionnaire | 5 minutes
  Improvement of low back pain measured by Oswestry Questionnaire: The results of the lumbar scale Oswestry disability percentage will be obtained. Results of the initial measurement, final month of treatment and compared.

SECONDARY OUTCOMES:
Centre of Pressure Displacement | 5 minutes
  Stabilometry used to assess Centre of Pressure Displacement. The stabilometric results will be obtained in percentages. The most important variables are the percentage of load anterior, load posterior, load right side and load left side.
  Results of the initial measurement, final month of treatment and compared.